CLINICAL TRIAL: NCT05120648
Title: Effects of Biofeedback on Somatic Symptoms, Psychological Adjustment and Health Status of UCLA Patients
Brief Title: Effects of Biofeedback on Somatic Symptoms
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Natacha D. Emerson, Assistant Clinical Professor, University of California, Los Angeles
Other Study IDs: 21-000741
Record Dates: First submitted 2021-09-13; First posted 2021-11-15 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Somatic Symptom
MeSH Terms: conditions — Medically Unexplained Symptoms | interventions — Biofeedback, Psychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate enrollment
  Interventions: Behavioral: Biofeedback
- Wait-list controls
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Behavioral: Biofeedback — We propose to study whether patients who complete a clinical six-session biofeedback protocol will demonstrate improvements in mental and physical health.

SUMMARY:
Biofeedback is a therapeutic paradigm that teaches patients how to gain awareness and control over previously unrecognized sympathetic changes such as body temperature, blood pressure, and heart rate. We propose to use a six session biofeedback protocol that includes heart-rate variability (HRV) biofeedback, respiration/relaxation training, and body temperature control to treat UCLA patients with chronic medical conditions (e.g. pulmonary, neurology) and somatic symptoms (pain, psychosomatic non-epileptic seizures, panic attacks, long-COVID symptoms). The aim of the study is to determine whether patients who complete a six-session biofeedback protocol report a decrease in somatic symptoms, and improvements in self-rated mental health (depression, anxiety, quality of life) after the program and at three-months follow-up. The investigators will also study whether these improvements are also related to reduced healthcare utilization.

DETAILED DESCRIPTION:
Biofeedback is a therapeutic paradigm that teaches patients how to gain awareness and control over previously unrecognized sympathetic changes such as body temperature, blood pressure, and heart rate. Through a series of mind-body techniques, patients are taught to reduce sympathetic responses, leading to self-regulation over physiological responses that affect somatic sensitivity. The investigators propose to use a six session biofeedback protocol that includes heart-rate variability (HRV) biofeedback, respiration/relaxation training, and body temperature control to treat UCLA patients with chronic medical conditions (e.g. pulmonary, neurology) and somatic symptoms (pain, psychosomatic non-epileptic seizures, panic attacks, long-COVID symptoms). The aim of the study is to determine whether patients who complete a six-session biofeedback protocol report a decrease in somatic symptoms, and improvements in self-rated mental health (depression, anxiety, quality of life) after the program and at three-months follow-up. The investigators will also study whether these improvements are also related to reduced healthcare utilization.

The investigators plan to recruit up to 100 participants in the study. Participants who are screened as eligible for biofeedback for their physical ailments or psychological complaints will be asked complete a set of questionnaires before, after, and three months' post-treatment to evaluate the utility of the biofeedback treatment protocol. These questionnaires will be available online and will be completed from home. Participants who are eligible to participate but cannot complete questionnaires from home will be given the option of completing the questionnaires in the office before the first biofeedback session. Participants that cannot be immediately enrolled in the protocol due to scheduling reasons will be asked to complete the questionnaires at recruitment to serve as wait-list controls. They will complete the same consent as other participants. The investigators anticipate that questionnaires will take 30 minutes to complete, totaling about 90 minutes for participants immediately enrolled and 120 minutes for wait-list controls.

Each biofeedback session will take 1 hour each. Session 1 of biofeedback will present the rationale and evidence for the treatment, teach breathing techniques, and introduce the biofeedback sensors for respiration, heart rate and temperature using the Biotrace software. The session will focus on breathing rate practice. Session 2 will introduce heart rate variability (HRV), cover breathing rhythm, and focus on the completion Resonance Frequency Assessment, an exercise to identify a participant's ideal breath rate for sustaining HRV. Session 3 will continue HRV practice using a separate software with video games, Alive. Session 4 will repeat session 3 but with more challenging practice of HRV video games. Session 5 will continue HRV practice in the first software (Biotrace) then will introduce participants to temperature control. Session 6 will repeat Session 5 but with more challenging practice for temperature control. Total time for participation will be approximately seven hours across three to six months.

ELIGIBILITY:
Inclusion Criteria:

* between 15-60 years of age
* English speaking
* minor participants must have one parent consent to research and treatment
* must have at least one qualifying somatic complaint (seizure-like spells, pain, nausea) or have psychosocial distress related to the management of their medical conditions (comorbid panic attacks, low mood, etc.).

Exclusion Criteria:

* severe psychopathology (e.g., psychosis, active suicidality, moderate to severe intellectual impairment).

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: (1) participants must be between 15-60; (2) English speaking; (3) minor participants must have one parent consent to research and treatment; (4) participants must have at least one qualifying somatic complaint (seizure-like spells, pain, nausea) or have psychosocial distress related to the management of their medical conditions (comorbid panic attacks, low mood, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in depression score on the PHQ-9 | 3 months and 6 months
  Improvement in self-rated depressive sx on the PHQ-9
Change in quality of life (QOL) | 3 months and 6 months
  Improvement in self-rated QOL on the SF-36
Change in anxiety | 3 months and 6 months
  Improvement in self-rated anxiety sx on the GAD-7
Reduced physical symptoms | 3 months and 6 months
  Improvement in self-rated physical symptoms on the PHQ-15
Improved self-efficacy | 3 months and 6 months
  Improvement in self-rated self-efficacy on the Self-efficacy for Managing Chronic Disease 6-item Scale
Reduced health anxiety | 3 months and 6 months
  Reduced scores on the self-reported Health Anxiety Inventory
Improved sleep | 3 months and 6 months
  Improved sleep and reduced insomnia on the PSQI

SECONDARY OUTCOMES:
Reduced healthcare utilization | 3 months and 6 months
  Fewer medical visits, hospitalizations, ER visits and use of prescription medications by self-report

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Emerson ND, Lavretsky H, Pittman WQ, Viswanathan N, Siddarth P. An open trial of biofeedback for long COVID. J Psychosom Res. 2024 Apr;179:111625. doi: 10.1016/j.jpsychores.2024.111625. Epub 2024 Feb 23. PMID 38458016